CLINICAL TRIAL: NCT06000670
Title: Efficacy of Autologous Adipose Derived Stromal Vascular Fraction for Musculoskeletal Conditions
Acronym: SVF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Amer Mansour, consultant orthopedic surgeon, Dubai Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DHA
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; knee chondromalacia
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Masking Description: investigator is blinded to clinical and radiological assessments .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- knee osteoarhritis (Experimental): patients with grade 2 and above chondromlacia as well as all grades of osteoarhtritis
  Interventions: Procedure: stromal vascular fraction injection in the osteoarthritic knee

INTERVENTIONS:
Procedure: stromal vascular fraction injection in the osteoarthritic knee — stromal vascular fraction harvested from mid abdominal wall under sedation and seperated from fat using mechanical centrifugation .injection of 5 cc of the SVF in the affected knee.

SUMMARY:
clinical efficacy of autologous stromal vascular fraction SVF,for inflammatory and degenerative conditions of the knees

DETAILED DESCRIPTION:
to evaluate the clinical effectiveness of point of care autologous adipose derived stromal vascular fraction (SVF) alone or in combination with exosomes,for inflammatory and degenerative conditions of the knees.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis any grade

  * knee chondromalacia grade 2 and above

Exclusion Criteria:

* active HIV
* pregnant women
* Mental disease
* severe cardio vascular disease
* severe coagulation disorders
* infected tissues
* patients on other experimental studies within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-12-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
change in pain level | 2 years
  visual analog scale 0-10 ( 10 being worst)

SECONDARY OUTCOMES:
percentage cartilage thickness change | 2 years
  as measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: DHA DHA, Study Director — dubai health autority

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: cell surgical network — https://stemcellrevolution.com/